CLINICAL TRIAL: NCT01196871
Title: An Open-label Phase 2A Study to Investigate Drug-Drug Interactions Between AT1001 (Migalastat Hydrochloride) and Agalsidase in Subjects With Fabry Disease
Brief Title: Drug-Drug Interaction Study Between AT1001 (Migalastat Hydrochloride) and Agalsidase in Participants With Fabry Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AT1001-013
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Fabry Disease
Keywords: Amicus Therapeutics; AT1001; Galafold; Migalastat; Pharmacokinetics
MeSH Terms: conditions — Fabry Disease | interventions — migalastat; larazotide acetate; agalsidase beta; agalsidase alfa

STUDY DESIGN:
Intervention Model Description: A 2-stage design was used to study the effects of 2 dose levels of migalastat, while a 2- or 3-period design within each stage enabled study of the effects of one drug on the PK, pharmacodynamics, and safety of the other drug.
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) (Experimental)
  Interventions: Drug: Migalastat HCl; Biological: Agalsidase Beta
- Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) (Experimental)
  Interventions: Drug: Migalastat HCl; Biological: Agalsidase Beta
- Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) (Experimental)
  Interventions: Drug: Migalastat HCl; Biological: Agalsidase Alfa
- Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) (Experimental)
  Interventions: Drug: Migalastat HCl; Biological: Agalsidase Beta
- Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) (Experimental)
  Interventions: Drug: Migalastat HCl; Biological: Agalsidase Beta
- Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg) (Experimental)
  Interventions: Drug: Migalastat HCl; Biological: Agalsidase Alfa

INTERVENTIONS:
Drug: Migalastat HCl — Oral capsules, single dose
  Other Names: AT1001; Galafold; migalastat
Biological: Agalsidase Beta — IV infusion, single dose
  Other Names: Fabrazyme
  Arms: Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg); Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg); Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg); Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg)
Biological: Agalsidase Alfa — IV infusion, single dose
  Other Names: Replagal
  Arms: Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg); Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)

SUMMARY:
The objective was to determine the effects of a single dose of migalastat hydrochloride (HCl) (migalastat) 150 and 450 milligrams (mg) on the safety and plasma pharmacokinetics (PK) of agalsidase and the effects of agalsidase on the safety and PK of migalastat 150 mg.

DETAILED DESCRIPTION:
This open-label study was conducted in 2 stages (Stage 1, Stage 2). Stage 1 included migalastat 150 mg; Stage 2 included migalastat 450 mg. Each dose of migalastat was selected to evaluate interaction with each of 3 doses of recombinant agalsidase: 0.5 mg/kilogram (kg) agalsidase beta; 1.0 mg/kg agalsidase beta; 0.2 mg/kg agalsidase alfa.

Migalastat was administered orally. Agalsidase alfa was administered as a 40-minute intravenous (IV) infusion and agalsidase beta was administered as a 2-hour (hr) IV infusion.

Stage 1 consisted of 3 treatment periods with 14 days intervening between each period.

Period 1, Day 1: agalsidase was administered alone.

Period 2, Day 1: migalastat was administered, followed 2 hrs later by agalsidase.

Period 3, Day 7: migalastat was administered alone.

Stage 2 consisted of two 14-day treatment periods in which the plasma exposure of migalastat was characterized when migalastat was administered with agalsidase solely to confirm the attainment of adequate migalastat plasma concentrations.

Period 1, Day 1: agalsidase was administered as an IV infusion using a calibrated infusion pump.

Period 2, Day 1: migalastat was administered, followed 2 hrs later by agalsidase.

ELIGIBILITY:
Inclusion Criteria:

* Male diagnosed with Fabry disease and between 18 and 65 years of age, inclusive
* Body mass index between 18-35 kg per meter squared
* Had initiated treatment with agalsidase at least 1 month prior to screening, and had received at least 2 infusions before screening
* Had stable dose level, dosing regimen, and form of agalsidase for at least 1 month before screening
* Had an estimated creatinine clearance greater than or equal to 50 milliliters (mL)/minute at screening
* Agreed to use medically accepted methods of contraception during the study and for 30 days after study completion
* Were willing and able to provide written informed consent

Exclusion Criteria:

* Had a documented transient ischemic attack, ischemic stroke, unstable angina, or myocardial infarction within the 3 months before screening
* Had clinically significant unstable cardiac disease (for example, cardiac disease requiring active management, such as symptomatic arrhythmia, unstable angina, or New York Heart Association class III or IV congestive heart failure)
* History of allergy or sensitivity to study drug (including excipients) or other iminosugars (such as miglustat, miglitol)
* Required a concomitant medication prohibited by the protocol: Glyset® (miglitol), or Zavesca® (miglustat)
* Any investigational/experimental drug or device within 30 days of screening, except for use of investigational enzyme replacement therapy for Fabry disease
* Had any intercurrent illness or condition that might have precluded the participant from fulfilling the protocol requirements or suggested to the investigator that the potential participant might have had an unacceptable risk by participating in this study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02-02 (Actual); Primary Completion 2012-10-09 (Actual); Study Completion 2012-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor Clinical Research, Study Director — Amicus Therapeutics
Locations (10):
- United States (5):
  - Birmingham, Alabama
  - Decatur, Georgia
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Springfield, Virginia
- Australia (2):
  - Nedlands
  - Parkville
- Edegem, Belgium
- Montreal, Canada
- Amsterdam, Netherlands

REFERENCES:
- [Result] Warnock DG, Bichet DG, Holida M, Goker-Alpan O, Nicholls K, Thomas M, Eyskens F, Shankar S, Adera M, Sitaraman S, Khanna R, Flanagan JJ, Wustman BA, Barth J, Barlow C, Valenzano KJ, Lockhart DJ, Boudes P, Johnson FK. Oral Migalastat HCl Leads to Greater Systemic Exposure and Tissue Levels of Active alpha-Galactosidase A in Fabry Patients when Co-Administered with Infused Agalsidase. PLoS One. 2015 Aug 7;10(8):e0134341. doi: 10.1371/journal.pone.0134341. eCollection 2015. PMID 26252393

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The total number of unique participants in this study was 20: 3 from Stage 1 were re-enrolled and newly identified in Stage 2. Of those, 1 initially received 0.5 milligrams (mg)/kilogram (kg) agalsidase beta; after resolution of an agalsidase beta shortage, their dose was increased to 1.0 mg/kg; all remaining visits were completed at this dose.
Groups:
- Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg): Stage 1: This arm consisted of 3 sequential treatment periods (Period 1 - Period 3). A single 150-mg oral dose (1 capsule) of migalastat hydrochloride (HCl) (migalastat) 2 hours (hr) before initiation of an intravenous (IV) infusion of 0.5 mg/kg mg/kg agalsidase beta.
- Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg): Stage 1: This arm consisted of 3 sequential treatment periods (Period 1 - Period 3). A single 150-mg oral dose (1 capsule) of migalastat HCl 2 hr before initiation of an IV infusion of 1.0 mg/kg agalsidase beta.
- Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg): Stage 1: This arm consisted of 3 sequential treatment periods (Period 1 - Period 3). A single 150-mg oral dose (1 capsule) of migalastat HCl 2 hr before initiation of an IV infusion of 0.2 mg/kg agalsidase alfa.
- Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg): Stage 2: This arm consisted of 2 sequential treatment periods (Period 1, Period 2). A single 450 mg oral dose (3 × 150-mg capsules) of migalastat HCl 2 hr before initiation of an IV infusion of 0.5 mg/kg agalsidase beta.
- Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg): Stage 2: This arm consisted of 2 sequential treatment periods (Period 1, Period 2). A single 450 mg oral dose (3 × 150-mg capsules) of migalastat HCl 2 hr before initiation of an IV infusion of 1.0 mg/kg agalsidase beta.
- Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg): Stage 2: This arm consisted of 2 sequential treatment periods (Period 1, Period 2). A single 450 mg oral dose (3 x 150-mg capsules) of migalastat HCl 2 hr before initiation of an IV infusion of 0.2 mg/kg agalsidase alfa.
Period: Stage 1: Period 1
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)
Started | 5 | 3 | 4 | 0 (Zero participants noted since these participants started in Stage 2) | 0 (Zero participants noted since these participants started in Stage 2) | 0 (Zero participants noted since these participants started in Stage 2)
PK Population (Participants with evaluable PK data who successfully completed at least Period 1 and 2 in any stage) | 5 | 3 | 4 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug (Safety Population) | 5 | 3 | 4 | 0 | 0 | 0
Completed | 5 | 3 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 1: Period 2
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)
Started | 5 | 3 | 4 | 0 (Zero participants noted since these participants started in Stage 2) | 0 (Zero participants noted since these participants started in Stage 2) | 0 (Zero participants noted since these participants started in Stage 2)
PK Population (Participants with evaluable PK data who successfully completed at least Period 1 and 2 in any stage) | 5 | 3 | 4 | 0 | 0 | 0
Completed | 5 | 3 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 1: Period 3
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)
Started | 5 | 3 | 4 | 0 (Zero participants noted since these participants started in Stage 2) | 0 (Zero participants noted since these participants started in Stage 2) | 0 (Zero participants noted since these participants started in Stage 2)
Completed | 5 | 3 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2: Period 1
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)
Started | 0 (Zero participants noted because participants had completed Stage 1) | 0 (Zero participants noted because participants had completed Stage 1) | 0 (Zero participants noted because participants had completed Stage 1) | 2 (Both participants re-enrolled into Stage 2 after completing Stage 1) | 5 (One participant re-enrolled into Stage 2 after completing Stage 1) | 4
Received at Least 1 Dose of Study Drug (Safety Population) | 0 | 0 | 0 | 2 | 5 | 4
PK Population (Participants with evaluable PK data who successfully completed at least Period 1 and 2 in any stage) | 0 | 0 | 0 | 1 | 5 | 4
Completed | 0 | 0 | 0 | 2 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2: Period 2
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)
Started | 0 (Zero participants noted because participants had completed Stage 1) | 0 (Zero participants noted because participants had completed Stage 1) | 0 (Zero participants noted because participants had completed Stage 1) | 1 (One participant switched agalsidase dose from 0.5 mg/kg in Period 1 to 1.0 mg/kg in Period 2) | 6 (One participant switched agalsidase dose from 0.5 mg/kg in Period 1 to 1.0 mg/kg in Period 2) | 4
PK Population (Participants with evaluable PK data who successfully completed at least Period 1 and 2 in any stage) | 0 | 0 | 0 | 1 | 6 | 4
Completed | 0 | 0 | 0 | 1 | 6 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: all participants who received at least 1 dose of agalsidase or migalastat. All safety analyses were performed using this set. Participants were analyzed according to treatment received. Three participants from Stage 1 were re-enrolled and newly identified in Stage 2, with 1 receiving both 0.5 and 1.0 mg/kg agalsidase beta.
Groups:
- Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg): Stage 1: This arm consisted of 3 sequential treatment periods (Period 1 - Period 3). A single 150-mg oral dose (1 capsule) of migalastat HCl 2 hr before initiation of an IV infusion of 0.5 mg/kg agalsidase beta.
- Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg): Stage 2: This arm consisted of 2 sequential treatment periods (Period 1, Period 2). A single 450-mg oral dose (3 × 150-mg capsules) of migalastat HCl 2 hr before initiation of an IV infusion of 0.5 mg/kg agalsidase beta.
- Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg): Stage 2: This arm consisted of 2 sequential treatment periods (Period 1, Period 2). A single 450-mg oral dose (3 × 150-mg capsules) of migalastat HCl 2 hr before initiation of an IV infusion of 1.0 mg/kg agalsidase beta.
- Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg): Stage 2: This arm consisted of 2 sequential treatment periods (Period 1, Period 2). A single 450-mg oral dose (3 x 150-mg capsules) of migalastat HCl 2 hr before initiation of an IV infusion of 0.2 mg/kg agalsidase alfa.
- Total: Total of all reporting groups
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg) | Total
Number analyzed (Participants) | 5 | 3 | 4 | 2 | 6 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The total number of unique participants in this study was 20: 3 from Stage 1 were re-enrolled and newly identified in Stage 2. The total number of participants in Stage 2 was 11. One participant received both 0.5 and 1.0 mg/kg agalsidase beta (450 mg migalastat) in Stage 2 and appears under both treatment groups.
  years
    Stage 1: number analyzed (Participants) | 5 | 3 | 4 | 0 | 0 | 0 | 12
    Stage 1 | 50.6 (6.88) | 45.7 (8.02) | 43.5 (5.07) |  |  |  | 47.0 (6.84)
    Stage 2: number analyzed (Participants) | 0 | 0 | 0 | 2 | 6 | 4 | 12
    Stage 2 |  |  |  | 53.5 (2.12) | 38.7 (12.16) | 38.5 (9.15) | 40.1 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The total number of unique participants in this study was 20: 3 from Stage 1 were re-enrolled and newly identified in Stage 2. The total number of participants in Stage 2 was 11. One participant received both 0.5 and 1.0 mg/kg agalsidase beta (450 mg migalastat) in Stage 2 and appears under both treatment groups.
  Participants
    Stage 1: number analyzed (Participants) | 5 | 3 | 4 | 0 | 0 | 0 | 12
    Stage 1: Female | 0 | 0 | 0 |  |  |  | 0
    Stage 1: Male | 5 | 3 | 4 |  |  |  | 12
    Stage 2: number analyzed (Participants) | 0 | 0 | 0 | 2 | 6 | 4 | 12
    Stage 2: Female |  |  |  | 0 | 0 | 0 | 0
    Stage 2: Male |  |  |  | 2 | 6 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change In Area Under The Plasma Concentration Versus Time Curve (AUC) For Active α-Galactosidase A (α-Gal A) Levels After Administration Of Migalastat
Description: This measure characterized the effects of migalastat on the plasma PK of agalsidase by measurement of the active α-Gal A enzyme level in plasma using a qualified assay that measured the rate of enzyme activity using an artificial, fluorescent substrate. The agalsidase plasma PK parameter values for AUC extrapolated from time 0 to infinity (AUCinfinity) and AUC to the last time point at which concentration is quantified (AUC0-t) are reported in hr*[nanomoles/hr/milliliter] (hr*[nmol/hr/mL]). In Period 1 of Stages 1 and 2, blood samples were collected: immediately before the agalsidase infusion and over a 24-hr period after infusion; on Days 2, 7, and 14. In Period 2 of Stages 1 and 2, blood samples were collected: prior to dosing with migalastat (2 hr prior to the agalsidase infusion) and 1 hr after migalastat dosing; immediately before initiation of the agalsidase infusion and over a 24-hr period after initiation of the agalsidase infusion; on Days 2, 7, and 14.
Time Frame: 0 hr, 2 hr, 2 days, 7 days, 14 days post dose
Population: PK Population: all participants with evaluable PK parameter data who had successfully completed at least Period 1 and Period 2 in any stage. All PK analyses were performed using the PK population.
Measure: Mean (Standard Deviation); unit: hr*[nmol/hr/mL]
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)
Number analyzed (Participants) | 5 | 3 | 4 | 1 | 6 | 4
hr*[nmol/hr/mL]
  Period 1: AUC0-t | 1132.72 (223.215) | 4730.47 (1045.068) | 384.20 (86.904) | 2409.02 (NA) — Single Participant: Statistical analysis not performed. | 5670.76 (3926.295) | 787.23 (509.967)
  Period 2: AUC0-t | 3255.09 (904.716) | 9541.21 (2813.139) | 1602.58 (425.798) | 6127.75 (NA) — Single Participant: Statistical analysis not performed. | 9908.56 (3097.746) | 2199.98 (875.140)
  Period 1: AUCinfinity | 1145.73 (217.894) | 4871.66 (1242.965) | 388.10 (83.770) | 2523.87 (NA) — Single Participant: Statistical analysis not performed. | 5851.62 (4345.407) | 800.38 (509.308)
  Period 2: AUCinfinity | 3287.09 (907.073) | 9765.04 (3118.875) | 1626.67 (407.595) | 6197.71 (NA) — Single Participant: Statistical analysis not performed. | 10280.79 (3399.342) | 2253.95 (859.586)
Statistical Analysis 1: Comparison: Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) vs Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) vs Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg); Statistical Analysis of Stage 1 AUC0-t Data: Point estimates for the geometric means and their 90% confidence interval (CI) are obtained by exponentiating the least squares mean and the lower and upper bounds of the 90% CI of the natural log-transformed data; Test type: Other — Geometric means for each treatment combination is obtained from the linear mixed effects model Log (parameter) = Intercept + ß*Treatment + Error; AUC0-t Ratio = 2.942, 90% CI 2-sided [2.439 to 3.548] — The ratios of the geometric means (combination/alone) and its 90% CI are obtained by exponentiating the least squares mean difference and its 90% CI of the natural log-transformed data
Statistical Analysis 2: Comparison: Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) vs Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) vs Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg); Statistical Analysis of Stage 1 AUCinfinity Data: Point estimates for the geometric means and their 90% CI are obtained by exponentiating the least squares mean and the lower and upper bounds of the 90% CI of the natural log-transformed data; Test type: Other — [test comment as in outcome 1, analysis 1]; AUCinfinity Ratio = 2.942, 90% CI 2-sided [2.431 to 3.560] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) vs Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) vs Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg); Statistical Analysis of Stage 2 AUC0-t Data: Point estimates for the geometric means and their 90% CI are obtained by exponentiating the least squares mean and the lower and upper bounds of the 90% CI of the natural log-transformed data; Test type: Other — [test comment as in outcome 1, analysis 1]; AUC0-t Ratio = 2.354, 90% CI 2-sided [1.826 to 3.035] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) vs Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) vs Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg); Statistical Analysis of Stage 2 AUCinfinity Data: Point estimates for the geometric means and their 90% CI are obtained by exponentiating the least squares mean and the lower and upper bounds of the 90% CI of the natural log-transformed data; Test type: Other — [test comment as in outcome 1, analysis 1]; AUCinfinity Ratio = 2.375, 90% CI 2-sided [1.839 to 3.068] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Change In Maximum Observed Plasma Concentration (Cmax) For Active α-Gal A Levels After Administration Of Migalastat
Description: This measure characterized the effects of migalastat on the plasma PK of agalsidase by measurement of the active α-Gal A enzyme level in plasma using a qualified assay that measured the rate of enzyme activity using an artificial, fluorescent substrate. The agalsidase plasma PK parameter value for Cmax is reported in nmol/hr/mL. In Period 1 of Stages 1 and 2, blood samples were collected: immediately before the agalsidase infusion and over a 24-hr period after infusion; on Days 2, 7, and 14. In Period 2 of Stages 1 and 2, blood samples were collected: prior to dosing with migalastat (2 hr prior to the agalsidase infusion) and 1 hr after migalastat dosing; immediately before initiation of the agalsidase infusion and over a 24-hr period after initiation of the agalsidase infusion; on Days 2, 7, and 14.
Time Frame: 0 hr, 2 hr, 2 days, 7 days, 14 days post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/hr/mL
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)
Number analyzed (Participants) | 5 | 3 | 4 | 1 | 6 | 4
nmol/hr/mL
  Period 1:Cmax | 514.18 (87.458) | 1682.13 (407.862) | 309.02 (91.568) | 684.36 (NA) — Single Participant: Statistical analysis not performed. | 1775.12 (684.734) | 370.91 (113.362)
  Period 2: Cmax | 899.93 (235.701) | 2400.86 (928.257) | 515.34 (77.207) | 1351.18 (NA) — Single Participant: Statistical analysis not performed. | 2413.31 (798.090) | 619.00 (141.411)
Statistical Analysis 1: Comparison: Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) vs Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) vs Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg); Statistical Analysis of Stage 1 Cmax Data: Point estimates for the geometric means and their 90% CI are obtained by exponentiating the least squares mean and the lower and upper bounds of the 90% CI of the natural log-transformed data; Test type: Other — [test comment as in outcome 1, analysis 1]; Cmax Ratio = 1.629, 90% CI 2-sided [1.440 to 1.843] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) vs Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) vs Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg); Statistical Analysis of Stage 2 Cmax Data: Point estimates for the geometric means and their 90% CI are obtained by exponentiating the least squares mean and the lower and upper bounds of the 90% CI of the natural log-transformed data; Test type: Other — [test comment as in outcome 1, analysis 1]; Cmax Ratio = 1.546, 90% CI 2-sided [1.300 to 1.838] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Change In Time To Maximum Observed Plasma Concentration (Tmax) And Terminal Elimination Half-life (T1/2) For Active α-Gal A Levels After Administration Of Migalastat
Description: This measure characterized the effects of migalastat on the plasma PK of agalsidase by measurement of the active α-Gal A enzyme level in plasma using a qualified assay that measured the rate of enzyme activity using an artificial, fluorescent substrate. The agalsidase plasma PK parameter values for tmax and t1/2 are reported in hr. In Period 1 of Stages 1 and 2, blood samples were collected: immediately before the agalsidase infusion and over a 24-hr period after infusion; on Days 2, 7, and 14. In Period 2 of Stages 1 and 2, blood samples were collected: prior to dosing with migalastat (2 hr prior to the agalsidase infusion) and 1 hr after migalastat dosing; immediately before initiation of the agalsidase infusion and over a 24-hr period after initiation of the agalsidase infusion; on Days 2, 7, and 14.
Time Frame: 0 hr, 2 hr, 2 days, 7 days, 14 days post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)
Number analyzed (Participants) | 5 | 3 | 4 | 1 | 6 | 4
hr
  Period 1: tmax | 2.07 (0.149) | 2.16 (0.778) | 0.75 (0.170) | 3.00 (NA) — Single Participant: Statistical analysis not performed. | 2.58 (0.801) | 0.75 (0.170)
  Period 2: tmax | 2.30 (0.447) | 2.41 (0.526) | 0.75 (0.170) | 3.00 (NA) — Single Participant: Statistical analysis not performed. | 2.58 (0.801) | 0.75 (0.170)
  Period 1: t1/2 | 3.91 (2.054) | 5.33 (4.082) | 4.48 (3.132) | 6.50 (NA) — Single Participant: Statistical analysis not performed. | 3.11 (1.875) | 5.15 (3.645)
  Period 2: t1/2 | 3.51 (1.304) | 4.30 (1.712) | 4.27 (1.536) | 3.49 (NA) — Single Participant: Statistical analysis not performed. | 4.96 (1.532) | 5.31 (2.462)

4. Primary Outcome: Change In AUC For Total α-Gal A Protein Levels After Administration Of Migalastat
Description: This measure characterized the effects of migalastat on the plasma PK of agalsidase by measurement of the α-Gal A protein level in plasma by Western blot using anti-human Gal A antibody. The agalsidase plasma PK parameter value for AUC0-t is reported in hr*[nanogram (ng)/hr/mL]. In Period 1 of Stages 1 and 2, blood samples were collected: immediately before the agalsidase infusion and over a 24-hr period after infusion; on Days 2, 7, and 14. In Period 2 of Stages 1 and 2, blood samples were collected: prior to dosing with migalastat (2 hr prior to the agalsidase infusion) and 1 hr after migalastat dosing; immediately before initiation of the agalsidase infusion and over a 24-hr period after initiation of the agalsidase infusion; on Days 2, 7, and 14.
Time Frame: 0 hr, 2 hr, 2 days, 7 days, 14 days post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*[ng/hr/mL]
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)
Number analyzed (Participants) | 5 | 3 | 4 | 1 | 6 | 4
hr*[ng/hr/mL]
  Period 1: AUC0-t | 57187.48 (47381.96) | 29905.87 (20470.28) | 42256.74 (13868.00) | 16229.13 (NA) — Single Participant: Statistical analysis not performed. | 17200.63 (16906.97) | 28770.37 (10941.44)
  Period 2: AUC0-t | 56895.40 (45753.77) | 34298.23 (17022.13) | 42528.55 (14652.93) | 16272.03 (NA) — Single Participant: Statistical analysis not performed. | 22031.50 (16754.04) | 29816.41 (8956.789)
Statistical Analysis 1: Comparison: Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) vs Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) vs Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg); Statistical Analysis of Stage 1 AUC0-t Data: Point estimates for the geometric means and their 90% CI are obtained by exponentiating the least squares mean and the lower and upper bounds of the 90% CI of the natural log-transformed data; Test type: Other — [test comment as in outcome 1, analysis 1]; AUC0-t Ratio = 1.025, 90% CI 2-sided [0.921 to 1.140] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) vs Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) vs Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg); [analysis description as in outcome 1, analysis 3]; Test type: Other — Geometric means for each treatment combination is obtained from the linear mixed effects mode Log (parameter) = Intercept + ß*Treatment + Error; AUC0-t Ratio = 1.256, 90% CI 2-sided [1.026 to 1.538] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Change In Percentage Of AUCinfinity Extrapolated From The Last Time Point At Which Concentration Is Quantified To Infinity (AUCextrapolated %) For Total α-Gal A Protein Levels After Administration Of Migalastat
Description: This measure characterized the effects of migalastat on the plasma PK of agalsidase by measurement of the α-Gal A protein level by Western blot using anti-human Gal A antibody. The agalsidase plasma PK parameter values for AUCextrapolated % are reported. AUCextrapolated % is reported instead of AUCinfinity because small but quantifiable concentrations of α-Gal A protein past 24 hr post-dose extrapolated to infinity comprised >50% of total AUC in most participants and were unevaluable. In Period 1 of Stages 1 and 2, blood samples were collected: immediately before the agalsidase infusion and over a 24-hr period after infusion; on Days 2, 7, and 14. In Period 2 of Stages 1 and 2, blood samples were collected: prior to dosing with migalastat (2 hr prior to the agalsidase infusion) and 1 hour after migalastat dosing; immediately before initiation of the agalsidase infusion and over a 24-hr period after initiation of the agalsidase infusion; on Days 2, 7, and 14.
Time Frame: 0 hr, 2 hr, 2 days, 7 days, 14 days post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of AUC
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)
Number analyzed (Participants) | 5 | 3 | 4 | 1 | 6 | 4
percentage of AUC
  Period 1 | 60.50 (22.241) | 27.55 (14.642) | 73.26 (13.324) | 8.49 (NA) — Single Participant: Statistical analysis not performed. | 12.30 (15.307) | 58.37 (11.065)
  Period 2 | 33.97 (31.662) | 17.91 (11.091) | 54.06 (21.538) | 3.25 (NA) — Single Participant: Statistical analysis not performed. | 11.90 (13.029) | 47.47 (18.832)

6. Primary Outcome: Change In Cmax For Total α-Gal A Protein Levels After Administration Of Migalastat
Description: This measure characterized the effects of migalastat on the plasma PK of agalsidase by measurement of the α-Gal A protein level in plasma by Western blot using anti-human Gal A antibody. The agalsidase plasma PK parameter values for Cmax is reported in nmol/hr/mL. In Period 1 of Stages 1 and 2, blood samples were collected: immediately before the agalsidase infusion and over a 24-hr period after infusion; on Days 2, 7, and 14. In Period 2 of Stages 1 and 2, blood samples were collected: prior to dosing with migalastat (2 hr prior to the agalsidase infusion) and 1 hr after migalastat dosing; immediately before initiation of the agalsidase infusion and over a 24-hr period after initiation of the agalsidase infusion; on Days 2, 7, and 14.
Time Frame: 0 hr, 2 hr, 2 days, 7 days, 14 days post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/hr/mL
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)
Number analyzed (Participants) | 5 | 3 | 4 | 1 | 6 | 4
nmol/hr/mL
  Period 1: Cmax | 7159.13 (4599.113) | 5156.74 (2411.601) | 3813.49 (1036.627) | 3141.84 (NA) — Single Participant: Statistical analysis not performed. | 3983.05 (1422.734) | 3587.46 (1181.299)
  Period 2: Cmax | 7060.29 (5016.147) | 5572.63 (1915.073) | 4196.18 (1264.763) | 2715.38 (NA) — Single Participant: Statistical analysis not performed. | 4170.15 (935.512) | 3773.21 (950.710)
Statistical Analysis 1: Comparison: Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) vs Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) vs Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg); [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Cmax Ratio = 1.034, 90% CI 2-sided [0.929 to 1.152] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) vs Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) vs Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg); [analysis description as in outcome 2, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 1]; Cmax Ratio = 1.063, 90% CI 2-sided [0.972 to 1.164] — [estimate comment as in outcome 1, analysis 1]

7. Primary Outcome: Change In Tmax And T1/2 For Total α-Gal A Protein Levels After Administration Of Migalastat
Description: This measure characterized the effects of migalastat on the plasma PK of agalsidase by measurement of the total α-Gal A protein level in plasma by Western blot using anti-human Gal A antibody. The agalsidase plasma PK parameter values for tmax and t1/2 are reported in hr. In Period 1 of Stages 1 and 2, blood samples were collected: immediately before the agalsidase infusion and over a 24-hr period after infusion; on Days 2, 7, and 14. In Period 2 of Stages 1 and 2, blood samples were collected: prior to dosing with migalastat (2 hr prior to the agalsidase infusion) and 1 hr after migalastat dosing; immediately before initiation of the agalsidase infusion and over a 24-hr period after initiation of the agalsidase infusion; on Days 2, 7, and 14.
Time Frame: 0 hr, 2 hr, 2 days, 7 days, 14 days post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)
Number analyzed (Participants) | 5 | 3 | 4 | 1 | 6 | 4
hr
  Period 1: tmax | 2.07 (0.149) | 2.16 (0.778) | 0.75 (0.170) | 3.00 (NA) — Single Participant: Statistical analysis not performed. | 2.50 (0.775) | 0.75 (0.170)
  Period 2: tmax | 2.10 (0.548) | 2.24 (0.750) | 0.75 (0.166) | 3.00 (NA) — Single Participant: Statistical analysis not performed. | 2.50 (0.548) | 0.75 (0.170)
  Period 1: t1/2 | 57.78 (40.019) | 17.77 (8.837) | 86.19 (92.048) | 2.96 (NA) — Single Participant: Statistical analysis not performed. | 6.71 (7.702) | 30.32 (5.010)
  Period 2: t1/2 | 23.10 (22.338) | 9.15 (5.621) | 32.95 (20.282) | 2.00 (NA) — Single Participant: Statistical analysis not performed. | 5.55 (5.553) | 28.05 (18.582)

8. Primary Outcome: Change In AUC For Migalastat After Administration Of Agalsidase
Description: This measure characterized the effects of agalsidase on the plasma PK of migalastat using a validated liquid chromatography-tandem mass spectrometry (LC-MS) assay. The migalastat plasma PK parameter values for AUCinfinity and AUC0-t are reported in hr*[ng/hr/mL]. In Period 2 of Stages 1 and 2, blood samples were collected: just before dosing with migalastat (2 hr prior to the agalsidase infusion) and at 1 hr after migalastat dosing; immediately before the agalsidase infusion and over a 24-hr period after infusion. In Period 3 (Stage 1 only), blood samples were collected before dosing and over the 24-hr period after administration of migalastat.
Time Frame: 0 hr, 1 day post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*[ng/hr/mL]
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)
Number analyzed (Participants) | 5 | 3 | 4 | 1 | 6 | 4
hr*[ng/hr/mL]
  Period 2: AUC0-t | 15717.87 (7140.484) | 9413.79 (2153.161) | 16051.81 (3441.663) | 49483.00 (NA) — Single Participant: Statistical analysis not performed. | 30450.61 (10750.31) | 33920.71 (8559.677)
  Period 3: AUC0-t | 13009.11 (3747.086) | 9285.71 (2270.875) | 16011.88 (5361.097) | NA (NA) — No Period 3 for Stage 2. | NA (NA) — No Period 3 for Stage 2. | NA (NA) — No Period 3 for Stage 2.
  Period 2: AUCinfinity | 15889.34 (7841.968) | 9653.09 (2185.031) | 16523.94 (3804.018) | 53034.59 (NA) — Single Participant: Statistical analysis not performed. | 31856.37 (11283.94) | 34700.89 (8429.954)
  Period 3: AUCinfinity | 13708.03 (4278.951) | 9597.10 (2253.444) | 16586.14 (5818.395) | NA (NA) — No Period 3 for Stage 2. | NA (NA) — No Period 3 for Stage 2. | NA (NA) — No Period 3 for Stage 2.
Statistical Analysis 1: Comparison: Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) vs Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) vs Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg); [analysis description as in outcome 4, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; AUC0-t Ratio = 1.059, 90% CI 2-sided [0.818 to 1.371] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) vs Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) vs Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg); [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 1]; AUCinfinity Ratio = 1.052, 90% CI 2-sided [0.807 to 1.371] — [estimate comment as in outcome 1, analysis 1]

9. Primary Outcome: Change In Cmax For Migalastat After Administration Of Agalsidase
Description: This measure characterized the effects of agalsidase on the plasma PK of migalastat using a validated liquid LC-MS assay. The migalastat plasma PK parameter values for Cmax are reported in nmol/hr/mL. In Period 2 of Stages 1 and 2, blood samples were collected: just before dosing with migalastat (2 hr prior to the agalsidase infusion) and at 1 hr after migalastat dosing; immediately before the agalsidase infusion and over a 24-hr period after infusion. In Period 3 (Stage 1 only), blood samples were collected before dosing and over the 24-hr period after administration of migalastat.
Time Frame: 0 hr, 1 day post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/hr/mL
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)
Number analyzed (Participants) | 5 | 3 | 4 | 1 | 6 | 4
nmol/hr/mL
  Period 2: Cmax | 1690.00 (606.548) | 1295.67 (501.654) | 2047.50 (192.592) | 4750.00 (NA) — Single Participant: Statistical analysis not performed. | 3763.33 (984.574) | 4455.00 (1840.697)
  Period 3: Cmax | 1634.00 (396.081) | 1374.00 (574.132) | 2035.00 (512.803) | NA (NA) — No Period 3 in Stage 2. | NA (NA) — No Period 3 in Stage 2. | NA (NA) — No Period 3 in Stage 2.
Statistical Analysis 1: Comparison: Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) vs Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) vs Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg); [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Cmax Ratio = 0.997, 90% CI 2-sided [0.791 to 1.259] — [estimate comment as in outcome 1, analysis 1]

10. Primary Outcome: Change In Tmax And T1/2 For Migalastat After Administration Of Agalsidase
Description: This measure characterized the effects of agalsidase on the plasma PK of migalastat using a validated LC-MS assay. The migalastat plasma PK parameter values for tmax and t1/2 are reported in hr. In Period 2 of Stages 1 and 2, blood samples were collected: just before dosing with migalastat (2 hr prior to the agalsidase infusion) and at 1 hr after migalastat dosing; immediately before the agalsidase infusion and over a 24-hr period after infusion. In Period 3 (Stage 1 only), blood samples were collected before dosing and over the 24-hr period after administration of migalastat.
Time Frame: 0 hr, 1 day post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)
Number analyzed (Participants) | 5 | 3 | 4 | 1 | 6 | 4
hr
  Period 2: tmax | 3.70 (0.651) | 3.33 (0.577) | 3.02 (0.818) | 4.00 (NA) — Single Participant: Statistical analysis not performed. | 3.33 (1.102) | 4.50 (1.000)
  Period 3: tmax | 3.03 (0.710) | 3.00 (0.000) | 3.03 (0.050) | NA (NA) — No Period 3 for Stage 2. | NA (NA) — No Period 3 for Stage 2. | NA (NA) — No Period 3 for Stage 2.
  Period 2: t1/2 | 5.39 (1.098) | 4.95 (0.335) | 4.86 (0.831) | 6.36 (NA) — Single Participant: Statistical analysis not performed. | 4.87 (1.202) | 4.44 (1.328)
  Period 3: t1/2 | 5.31 (1.241) | 5.05 (0.558) | 4.81 (0.601) | NA (NA) — No Period 3 for Stage 2. | NA (NA) — No Period 3 for Stage 2. | NA (NA) — No Period 3 for Stage 2.

11. Secondary Outcome: Change From Baseline To Day 7 In Active α-Gal A In Skin Following Treatment With Agalsidase Alone And Co-administration With Migalastat
Description: This measure characterized the effects of agalsidase and migalastat on α-Gal A activity in the skin using a qualified assay that measured the rate of enzyme activity using an artificial, fluorescent substrate. Baseline was defined as Day 1/Period 1 pre-infusion level. α-Gal A activity is reported in picomoles/mg/hr (pmol/mg/hr). Biopsy samples were obtained: on Day -1/Period 1; 24 hr after initiation of the infusion during Period 1 and Period 2; on Day 7 of Period 1 and Period 2.
Time Frame: Baseline, Day 7
Population: as for outcome 1
Measure: Mean (Full Range); unit: pmol/mg/hr
Arm/Group | Agalsidase Beta (0.5 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (150 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (150 mg) | Agalsidase Beta (0.5 mg/kg)-Migalastat (450 mg) | Agalsidase Beta (1.0 mg/kg)-Migalastat (450 mg) | Agalsidase Alfa (0.2 mg/kg)-Migalastat (450 mg)
Number analyzed (Participants) | 5 | 3 | 4 | 1 | 6 | 4
pmol/mg/hr
  Period 1: Day 2: number analyzed (Participants) | 5 | 2 | 3 | 1 | 6 | 1
  Period 1: Day 2 | 334 [-141 to 998] | 857 [795 to 919] | 121 [-52 to 371] | 89 [NA to NA] — Single Participant: Statistical analysis not performed. | 1936 [884 to 3162] | 18 [NA to NA] — Single Participant: Statistical analysis not performed.
  Period 2: Day 2: number analyzed (Participants) | 4 | 1 | 3 | 1 | 6 | 1
  Period 2: Day 2 | 1508 [221 to 4103] | 2977 [NA to NA] — Single Participant: Statistical analysis not performed. | 437 [35 to 1146] | 647 [NA to NA] — Single Participant: Statistical analysis not performed. | 4019 [1777 to 6168] | 160 [NA to NA] — Single Participant: Statistical analysis not performed.
  Period 1: Day 7: number analyzed (Participants) | 5 | 2 | 2 | 1 | 6 | 0
  Period 1: Day 7 | 137 [45 to 234] | 553 [315 to 791] | 139 [50 to 229] | 72 [NA to NA] — Single Participant: Statistical analysis not performed. | 613 [252 to 2001] |
  Period 2: Day 7: number analyzed (Participants) | 5 | 2 | 3 | 1 | 6 | 1
  Period 2: Day 7 | 574 [-200 to 2588] | 855 [460 to 1250] | 228 [11 to 606] | 235 [NA to NA] — Single Participant: Statistical analysis not performed. | 789 [-174 to 1935] | -100 [NA to NA] — Single Participant: Statistical analysis not performed.

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were monitored up to 5.5 months after the first dose of study drug. For Period (Pd) 1 and 2 of Stages 1 and 2, AEs were reported starting 1 day prior (Day -1) to the first dose of study drug (Agalsidase Beta [Agal-B] or Agalsidase Alfa [Agal-A]) to 1 month after the last dose of study drug. For Pd 3 of Stage 1, AEs were reported starting on the day of the first dose of study drug (Day 1) to 1 month after the last dose of study drug (Migalastat [Mig]).
Groups:
- Stage 1 Pd 1: 0.5 mg/kg Agal-B (Arm 1): Period 1 of Stage 1 consisted of IV administration of 0.5 mg/kg agalsidase beta.
- Stage 1 Pd 2: 150 mg Mig Before 0.5 mg/kg Agal-B (Arm 1): Period 2 of Stage 1 consisted of administration of a single 150-mg oral dose of migalastat HCl 2 hr before initiation of an IV infusion of 0.5 mg/kg agalsidase beta.
- Stage 1 Pd 3: 150 mg Mig (Arm 1); Stage 1 Pd 3: 150 mg Mig (Arm 2); Stage 1 Pd 3: 150 mg Mig (Arm 3): Period 3 of Stage 1 consisted of a single 150-mg oral dose of migalastat HCl.
- Stage 1 Pd 1: 1.0 mg/kg Agal-B (Arm 2): Period 1 of Stage 1 consisted of IV administration of 1.0 mg/kg agalsidase beta.
- Stage 1 Pd 2: 150 mg Mig Before 1.0 mg/kg Agal-B (Arm 2): Period 2 of Stage 1 consisted of administration of a single 150-mg oral dose of migalastat HCl 2 hr before initiation of an IV infusion of 1.0 mg/kg agalsidase beta.
- Stage 1 Pd 1: 0.2 mg/kg Agal-A (Arm 3): Period 1 of Stage 1 consisted of IV administration of 0.2 mg/kg agalsidase alfa.
- Stage 1 Pd 2: 150 mg Mig Before 0.2 mg/kg Agal-A (Arm 3): Period 2 of Stage 1 consisted of administration a single 150-mg oral dose of migalastat HCl 2 hr before initiation of an IV infusion of 0.2 mg/kg agalsidase alfa.
- Stage 2 Pd 1: 0.5 mg/kg Agal-B (Arm 4); Stage 2 Pd 1: 1.0 mg/kg Agal-B (Arm 5): Period 1 of Stage 2 consisted of IV administration of 0.5 mg/kg agalsidase beta.
- Stage 2 Pd 2: 450 mg Mig Before 0.5 mg/kg Agal-B (Arm 4): Period 2 of Stage 2 consisted of a single 450-mg oral dose (3 x 150-mg capsules) of migalastat HCl 2 hr before IV administration of 0.5 mg/kg agalsidase beta.
- Stage 2 Pd 2: 450 Mig Before 1.0 mg/kg Agal-B (Arm 5): Period 2 of Stage 2 consisted of a single 450-mg oral dose (3 x 150-mg capsules) of migalastat HCl 2 hr before IV administration of 1.0 mg/kg agalsidase beta.
- Stage 2 Pd 1: 0.2 mg/kg Agal-A (Arm 6): Period 1 of Stage 2 consisted of IV administration of 0.2 mg/kg agalsidase alfa.
- Stage 2 Pd 2: 450 Mig Before 0.2 mg/kg Agal-A (Arm 6): Period 2 of Stage 2 consisted of a single 450-mg oral dose (3 x 150-mg capsules) of migalastat HCl 2 hr before IV administration of 0.2 mg/kg agalsidase alfa.
Arm/Group | Stage 1 Pd 1: 0.5 mg/kg Agal-B (Arm 1) | Stage 1 Pd 2: 150 mg Mig Before 0.5 mg/kg Agal-B (Arm 1) | Stage 1 Pd 3: 150 mg Mig (Arm 1) | Stage 1 Pd 1: 1.0 mg/kg Agal-B (Arm 2) | Stage 1 Pd 2: 150 mg Mig Before 1.0 mg/kg Agal-B (Arm 2) | Stage 1 Pd 3: 150 mg Mig (Arm 2) | Stage 1 Pd 1: 0.2 mg/kg Agal-A (Arm 3) | Stage 1 Pd 2: 150 mg Mig Before 0.2 mg/kg Agal-A (Arm 3) | Stage 1 Pd 3: 150 mg Mig (Arm 3) | Stage 2 Pd 1: 0.5 mg/kg Agal-B (Arm 4) | Stage 2 Pd 2: 450 mg Mig Before 0.5 mg/kg Agal-B (Arm 4) | Stage 2 Pd 1: 1.0 mg/kg Agal-B (Arm 5) | Stage 2 Pd 2: 450 Mig Before 1.0 mg/kg Agal-B (Arm 5) | Stage 2 Pd 1: 0.2 mg/kg Agal-A (Arm 6) | Stage 2 Pd 2: 450 Mig Before 0.2 mg/kg Agal-A (Arm 6)
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/3 | 0/3 | 0/3 | 0/4 | 0/4 | 0/4 | 1/2 | 0/1 | 0/6 | 0/6 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/5 | 0/5 | 3/5 | 3/3 | 2/3 | 0/3 | 1/4 | 0/4 | 2/4 | 1/2 | 0/1 | 1/6 | 1/6 | 3/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 Pd 1: 0.5 mg/kg Agal-B (Arm 1) (N=5) | Stage 1 Pd 2: 150 mg Mig Before 0.5 mg/kg Agal-B (Arm 1) (N=5) | Stage 1 Pd 3: 150 mg Mig (Arm 1) (N=5) | Stage 1 Pd 1: 1.0 mg/kg Agal-B (Arm 2) (N=3) | Stage 1 Pd 2: 150 mg Mig Before 1.0 mg/kg Agal-B (Arm 2) (N=3) | Stage 1 Pd 3: 150 mg Mig (Arm 2) (N=3) | Stage 1 Pd 1: 0.2 mg/kg Agal-A (Arm 3) (N=4) | Stage 1 Pd 2: 150 mg Mig Before 0.2 mg/kg Agal-A (Arm 3) (N=4) | Stage 1 Pd 3: 150 mg Mig (Arm 3) (N=4) | Stage 2 Pd 1: 0.5 mg/kg Agal-B (Arm 4) (N=2) | Stage 2 Pd 2: 450 mg Mig Before 0.5 mg/kg Agal-B (Arm 4) (N=1) | Stage 2 Pd 1: 1.0 mg/kg Agal-B (Arm 5) (N=6) | Stage 2 Pd 2: 450 Mig Before 1.0 mg/kg Agal-B (Arm 5) (N=6) | Stage 2 Pd 1: 0.2 mg/kg Agal-A (Arm 6) (N=4) | Stage 2 Pd 2: 450 Mig Before 0.2 mg/kg Agal-A (Arm 6) (N=4)
Acroparaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 Pd 1: 0.5 mg/kg Agal-B (Arm 1) (N=5) | Stage 1 Pd 2: 150 mg Mig Before 0.5 mg/kg Agal-B (Arm 1) (N=5) | Stage 1 Pd 3: 150 mg Mig (Arm 1) (N=5) | Stage 1 Pd 1: 1.0 mg/kg Agal-B (Arm 2) (N=3) | Stage 1 Pd 2: 150 mg Mig Before 1.0 mg/kg Agal-B (Arm 2) (N=3) | Stage 1 Pd 3: 150 mg Mig (Arm 2) (N=3) | Stage 1 Pd 1: 0.2 mg/kg Agal-A (Arm 3) (N=4) | Stage 1 Pd 2: 150 mg Mig Before 0.2 mg/kg Agal-A (Arm 3) (N=4) | Stage 1 Pd 3: 150 mg Mig (Arm 3) (N=4) | Stage 2 Pd 1: 0.5 mg/kg Agal-B (Arm 4) (N=2) | Stage 2 Pd 2: 450 mg Mig Before 0.5 mg/kg Agal-B (Arm 4) (N=1) | Stage 2 Pd 1: 1.0 mg/kg Agal-B (Arm 5) (N=6) | Stage 2 Pd 2: 450 Mig Before 1.0 mg/kg Agal-B (Arm 5) (N=6) | Stage 2 Pd 1: 0.2 mg/kg Agal-A (Arm 6) (N=4) | Stage 2 Pd 2: 450 Mig Before 0.2 mg/kg Agal-A (Arm 6) (N=4)
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear canal erythema (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Faeces pale (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart sounds abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node palpable (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tinea capitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amaurosis fugax (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Incision site blister (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fabry's disease (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can only publish the results from this trial provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review. If requested, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication for an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.